CLINICAL TRIAL: NCT07019740
Title: Evaluatıon of sympathetıc Nervous System fındıngs and theır relatıonshıp wıth Symptoms ın patıents wıth Breast Cancer Related Lymphedema
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU.FTR.N.T.
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema, Breast Cancer
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Diagnosis-Related Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CASE GROUP: BREAST CANCER RELATED LYPMHEDEMA
  Interventions: Other: CASE GROUP
- CONTROL GROUP: HEALTHY GROUP
  Interventions: Other: CASE GROUP

INTERVENTIONS:
Other: CASE GROUP — SYMPATHETIC SKIN RESPONSE, CUTANEOUS QUIET PERIOD AND COMPASS-31 QUESTIONNAIRE EVALUATED

SUMMARY:
The aim of this study was to evaluate the sympathetic nervous system, small fiber functions and autonomic symptoms in patients with breast cancer related lymphedema and to investigate the relationship between these findings and patients' symptoms.

DETAILED DESCRIPTION:
This observational cross-sectional study aims to evaluate sympathetic nervous system activity, small fiber function, and autonomic symptoms in patients with breast cancer related lymphedema.

Electrophysiological parameters, including Sympathetic Skin Response (SSR) and Cutaneous Silent Period (CSP), will be recorded from both the affected and unaffected limbs using standardized neurophysiological techniques. Additionally, autonomic symptoms will be assessed using the Composite Autonomic Symptom Score 31 (COMPASS-31), and the impact of lymphedema on daily life will be evaluated with the Lymphedema Life Impact Scale (LLIS).

The study hypothesizes that sympathetic dysfunction and small fiber involvement may contribute to the pathophysiology of lymphedema and correlate with subjective symptoms such as pain, heaviness, and tightness.

Findings from this study are expected to provide insights into the potential role of the autonomic nervous system in breast cancer-related lymphedema and may support future consideration of sympathetic nervous system-targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient age group between 18-75 years
* To have been diagnosed with breast cancer-related lymphedema by imaging and/or clinical diagnostic methods

Exclusion Criteria:

History of upper extremity lymphedema due to causes other than breast cancer

* Lymphedema in other body parts
* Diagnosis of polyneuropathy or entrapment neuropathy in the upper extremity
* Presence of active infection at the assessment site
* Presence of congenital or acquired malformations at the evaluation site
* Those with any medical condition that may cause edema, such as severe heart or kidney failure

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: BREAST CANCER RELATED LYMPHEDEMA
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
SSR latency in affected and unaffected arms of patient with breast cancer related lymphedema | Day 1
  Sympathetic skin response (SSR) latency will be recorded bilaterally using standard surface electrodes placed on the palm and dorsum of the hand. Electrical stimulation will be applied to the median nerve at the wrist with parameters of 20-30 mA and 0.2 ms pulse duration. Latency is defined as the time between stimulus and onset of the first deflection in the recording and will be expressed in milliseconds.
SSR amplitude in affected and unaffected arms of patients with breast cancer related lymphedema | Day 1
  SSR amplitude will be recorded bilaterally using surface electrodes. Amplitude is measured as the peak-to-peak voltage of the waveform following stimulation of the median nerve at the wrist using standard stimulation parameters. Recordings will be performed with a standard EMG device and values will be reported in microvolts.
CSP latency in affected and unaffected arms pf patients with breast cancer related lymphedema | Day 1
  Cutaneous Silent Period (CSP) latency will be measured by applying painful electrical stimulation to the index finger and recording EMG activity from the abductor pollicis brevis muscle. Latency is defined as the time between the stimulus and the onset of EMG suppression. Standard protocols for CSP measurement will be followed.
CSP duration in affected and unaffected arms of patients with breast cancer related lymphedema | Day 1
  CSP duration will be calculated as the time between the onset of EMG suppression and the return to baseline voluntary EMG activity following electrical stimulation. Recordings will be made using an EMG system and reported in milliseconds.
COMPASS-31 total score and subdomains in patients with breast cancer related lymphedema | Day 1
  The Composite Autonomic Symptom Score 31 (COMPASS-31) questionnaire will be used to evaluate autonomic symptoms. It includes domains such as orthostatic intolerance, secretomotor, vasomotor, gastrointestinal, bladder, and pupillomotor symptoms. The total score ranges from 0 to 100, where higher scores indicate more severe autonomic dysfunction.

SECONDARY OUTCOMES:
Comparison of primary measurements with Lymphedema Life Impact Scale total score and subdomains in patients with breast cancer related lymphedema | Day 1
  The Lymphedema Life Impact Scale (LLIS) will be used to evaluate the impact of lymphedema on function, symptoms, and emotional well-being. Each item on the LLIS is scored using a 5-point likert scale, ranging from 1 to 5. Higher LLIS scores indicated greater disability and reduced quality of life in patients with breast cancer related lymphedemaParticipants will complete the questionnaire and scores will be correlated with electrophysiological and autonomic findings.
Comparison of primary measurements with limb volume difference between arms in patients with breast cancer related lymphedema | Day 1
  The volume of the affected and unaffected limbs will be calculated using a circumferential measurement method. Measurements will be taken at regular intervals along the limb, and limb volume will be estimated using the truncated cone formula:
  V = Σ [π × h × (C₁² + C₁×C₂ + C₂²) / 12π] where C₁ and C₂ are the circumferences at two adjacent levels and h is the distance between them. This approach allows for volume estimation without the use of water displacement. The interlimb volume difference (affected minus unaffected arm) will be calculated in milliliters and compared with primary outcome measures.
Comparison of primary measurements with pain rating in the affected arm in patients with breast cancer related lymphedema | Day 1
  Patients will rate their pain in the affected arm using a numeric rating scale from 0 (no pain) to 10 (worst pain imaginable). Scores will be compared with primary outcome measures.
Comparison of primary measurements with heaviness rating in the affected arm in patients with breast cancer related lymphedema | Day 1
  Patients will report their perception of heaviness in the affected arm using a numeric scale ranging from 0 to 10. These scores will be compared with SSR, CSP and Compass 31 results.
Comparison of primary measurements with tightness rating in the affected arm in patients with breast cancer related lymphedema | Day 1
  Patients will evaluate the tightness sensation in the affected limb on a 0-10 numeric rating scale. Data will be analyzed in association with SSR, CSP and Compass 31 results.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No